CLINICAL TRIAL: NCT02478658
Title: Circulatory Levels of Irisin in Response to Acute Resistance Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 504792A
Record Dates: First submitted 2015-02-03; First posted 2015-06-23 (Estimated); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Healthy
Keywords: irisin; resistance training; physical fitness; Volunteers
MeSH Terms: interventions — Exercise

ARMS (2):
- Intervention (Experimental): The acute intervention will consist of 1 session of training following the program:
  Resistance Training Exercises. Each participant in the intervention group will perform resistance-training exercises in the form of a circuit. The circuit will consist of 10 repetitions per exercise of 7 exercises: leg press, bent-over row, bench press, squats, dumbbell jump squats with raises, dead-lifts and weighted abdominal crunches, with approximately 30 sec of rest in between each exercise (based on the estimated time needed to move from one position to the next). Initial intensity 6-7 of RPE and ending the set at 9-10. Each participant will move through the circuit 3 times, with 2 to 3 minutes of rest between each round.
  Interventions: Other: exercise training
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: exercise training — high-intensity resistance training
  Arms: Intervention

SUMMARY:
Study the circulatory levels of irisin in response to one session of high-intensity resistance training in a group of healthy subjects.

DETAILED DESCRIPTION:
Objective: The purpose of this study is to study the circulating levels of irisin in response to acute high-intensity resistance training in a group of healthy young adults.

Sample: The sample will be comprised of adult men and women unpaid volunteers between the ages of 18 and 30. We will recruit 44 participants.

Pre- screening assessments: Informed consent, PAR-Q, Medical History and Exercise History will be used to determine health status and prior exercise experience. Menstrual cycle log will be required for female participants.

Pre-Intervention assessments (baseline):

* Anthropometric measurements and Body Composition: Height, triceps, thigh and calf skinfolds, biceps, thigh, hip, waist, and calf circumferences will be measured. Dual-energy x-ray absorptiometry (DEXA) will be performed to obtain body composition.
* Blood-related variables. Baseline glucose, lactate and hematocrit will be obtained from all participants prior to intervention. Lactate and Hematocrit will be obtained pre-intervention and post-intervention, and within 1 min post workout.

Irisin will be obtained from blood samples at baseline, during and after the training session. Irisin will be measured via a commercial enzyme-linked immunosorbent assay.

* Cardiopulmonary and Strength Fitness Testing. Cardiopulmonary fitness will be determined via maximum oxygen consumption testing. One maximum repetition (1-RM) will be used to assess the muscular fitness.
* Dietary Controls. Each participant will complete the Food Preference Questionnaire. In addition, the Automated Self-Administered 24-hour Recall (ASA24) will be collected for the day prior to the session.
* Familiarization. Participant will be instructed on the muscle conditioning techniques used for strength training so that the techniques can be mastered. The rate of perceived exertion (RPE) scale will also be used for familiarization during these sessions.
* Spontaneous Physical Activity: Daily activity level for 7 days will be collected.

Intervention: Resistance training will consist on a circuit training of 3 sets of 7 exercises focused on major muscle groups. Ten repetitions on each circuit at 70% of the maximum capacity will be performed. Acute intervention will consist of one session. Blood will be collected pre-session, at 45 min during the session, and immediately after the acute intervention exposure (post-session).

ELIGIBILITY:
Inclusion Criteria:

* Participants between 18 and 30 years old
* Males and Females
* Healthy

Exclusion Criteria:

* Participants with known health problems such as cardiovascular, pulmonary or metabolic disease will be excluded.
* Pregnant females will be excluded from the study.
* Any adults found taking medications that affect endocrine or cardiovascular function will also be excluded from the study.
* Individuals found to be less than 110 pounds will also be excluded due to the collection of blood during this study.
* Participants that exercise more than three times per week or strength train more than twice per week will be excluded.
* Individuals that have poor venous access or have expressed a fear of needles or having blood taken will also be excluded.
* Cigarette smoking (current or those who quit within the previous 6 months
* Hypertension
* Overweight and obese
* Pre-diabetics

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-02; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Serum irisin levels | 1 day
  Changes in irisin levels baseline, 45 min (during the training session), and post-training session

SECONDARY OUTCOMES:
Body composition assessment, as measured by DEXA and anthropometry | 1 day
  Body composition at baseline prior to the training session
Lactate levels | 1 day
  Intensity of exercise at the end of the session (post-training session)
Physical Fitness levels as measured by 1 RM (repetition maximum) and Cardio-respiratory maximal test | 1day
  Physical Fitness levels at baseline prior to the training session
Blood Glucose levels | 1 session (1 day)
  Blood Glucose levels at baseline prior to the training session
Diet assessment: 24 hour recall and Food Preference Questionnaire | 1day
  Dietary habits at baseline prior to the training session
Hematocrit concentration | 1 day
  Hematocrit levels at baseline and post-training session
Physical Activity assessment, as measured by Accelerometry. | 1 week
  Quantification of baseline Physical Activity levels at baseline prior to the training session

CONTACTS AND LOCATIONS:
Overall Officials: Maria Fernandez del Valle, PhD, Principal Investigator — Texas Tech University
Locations (1):
- Exercise and Sport Sciences Building, Lubbock, Texas, United States